CLINICAL TRIAL: NCT04266379
Title: A Randomized Clinical Trial to Assess the Efficacy of Adjunctive Closed Loop Control Versus Sensor and Pump Therapy in the Management of Type 1 Diabetes Prone to Hypoglycemia
Brief Title: Efficacy of Closed-loop Insulin Therapy in Adults Prone to Hypoglycemia
Acronym: DCLP2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Tandem Diabetes Care, Inc. (Industry); DexCom, Inc. (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL19_0351-(7826); 2019-A01906-51 (Registry Identifier: IDRCB); CIV-FR-19-12-031026 (Registry Identifier: EUDAMED); UC4DK108483 (NIH)
Record Dates: First submitted 2020-02-03; First posted 2020-02-12 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Type 1 Diabetes Mellitus With Hypoglycemia
Keywords: Type 1 diabetes; Hypoglycemia; Closed-loop insulin infusion
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Pancreas, Artificial; Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Closed-Loop Control (CLC) (Experimental): Closed-loop subcutaneous insulin infusion driven by continuous glucose monitoring through an algorithm
  Interventions: Device: Closed-loop insulin infusion driven by continuous glucose monitoring through an algorithm, in free-life conditions
- Sensor Augmented Pump (SAP) (Active Comparator): Closed-loop subcutaneous insulin infusion and continuous glucose monitoring manage by patient
  Interventions: Device: Continuous Subcutaneous Insulin Infusion and Continuous Glucose Monitoring

INTERVENTIONS:
Device: Closed-loop insulin infusion driven by continuous glucose monitoring through an algorithm, in free-life conditions — Continuous subcutaneous insulin infusion according to an automated algorithm from continuous glucose monitoring data
  Other Names: Artificial Pancreas
  Arms: Closed-Loop Control (CLC)
Device: Continuous Subcutaneous Insulin Infusion and Continuous Glucose Monitoring — Insulin delivered subcutaneously by a pump and manage by the patient with the help of a CGM sensor
  Other Names: Sensor Augmented Pump; CSII and CGM
  Arms: Sensor Augmented Pump (SAP)

SUMMARY:
This study is a RCT of 3 month at home comparing closed-loop control (CLC) system vs sensor and pump therapy (S&P), with a 3-month extension phase, in Type 1 diabetic patient prone to hypoglycemia. After a 2-week run-in phase with blinded CGM, patients who spent 5% or more time below 70mg/dL will be eligible to continue. They will will be randomly assigned 2:1 to the use of closed-loop control (CLC) using Tandem Control-IQ vs S&P for 3 months, which is the timing of the primary outcome for the RCT. After 3 months, the S&P group will use CLC for up to 3 months and the CLC group will continue using CLC for up to 3 additional months.

DETAILED DESCRIPTION:
This study is randomized controlled trial of 3 month at home closed-loop control (CLC) system vs sensor and pump therapy (S&P), with a 3-month extension phase. The objective is to assess the efficacy and safety of home use of a Control-to-Range (CTR) closed-loop (CL) system in patients with type 1 diabetes prone to hypoglycemia.

The CLC system will consist of Tandem Control-IQ Automated Insulin Delivery System (AIDS), including Tandem X2 insulin pump with embedded Control-IQ algorithm and Dexcom G6 CGM

After consent is signed, eligibility will be assessed. All participants will initiate a run-in phase of 2 weeks of blinded Dexcom G6 CGM wear and personal insulin pump.

Prior to overall initiation of the RCT, the time spent with CGM below 70 mg/dl during the run-in phase will be assessed. Only patients showing % time with CGM <70 mg/dl of 5% or above can be randomized. Included patients who cannot be randomized will be replaced.

Subsequent participants who show randomization criteria during the run-in phase will be randomly assigned 2:1 to the use of closed-loop control (CLC) using Tandem Control-IQ vs S&P for 3 months, which is the timing of the primary outcome for the RCT.

After 3 months, the S&P group will use CLC for up to 3 months and the CLC group will continue using CLC for up to 3 additional months.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year and using insulin for at least 1 year
2. Use of an insulin pump for at least 6 months
3. Age ≥18 .0 years old
4. HbA1c level <10.5% at screening
5. Clarke score >3 and/or experience of severe hypoglycemia during the previous 6 months
6. For females, not currently known to be pregnant If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all premenopausal women who are not surgically sterile. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
7. Willingness not to use glucose-lowering agents (such as Pramlintide, Metformin, GLP-1 analogs, SGLT2 inhibitors) during the study. This does not concern treatment with Metformin active and stable for more than 3 months prior the inclusion. Moreover, the use of SGLT2 inhibitors is not allowed in the 3 months prior to enrollment.
8. Willingness to suspend use of any personal CGM for the duration of the clinical trial
9. Willingness to establish network connectivity on at least a weekly basis
10. Currently using no insulins other than one of the following rapid-acting insulins at the time of enrollment: insulin lispro (Humalog), insulin aspart (Novolog). Patients using glulisine (Apidra) may switch to lispro or aspart at least one month prior to enrollment.
11. Investigator has confidence that the participant can successfully operate all study devices and is capable of adhering to the protocol
12. Subject is covered by social health or similar insurance
13. Informed consent form signed

Exclusion Criteria:

1. Use of SGLT2 inhibitors in the 3 months prior to enrollment
2. Hemophilia or any other bleeding disorder
3. A condition, which in the opinion of the investigator or designee, would put the participant or study at risk
4. Participation in another pharmaceutical or device trial at the time of enrollment or during the study
5. Employed by, or having immediate family members employed by Tandem or Dexcom
6. Persons deprived of freedom, protected by law or vulnerable persons
7. Any associated chronic disease or therapy (except insulin) affecting glucose metabolism
8. Impaired renal function (Creatinine Clearance < 30 ml/min)
9. Patient who had pancreas transplantation or pancreatic islet transplantation
10. Patient having severe problems of uncorrected hearing and/or visual acuity
11. Subjects with known allergy to CGM adhesives
12. Patients that have frequent exposure to magnetic resonance imaging (MRI), computed tomography (CT) scan, or high-frequency electrical heat (diathermy) treatment
13. Patient without any social or familial support able to intervene in case of severe hypoglycemic episode

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-05-13 (Actual); Primary Completion 2022-11-03 (Estimated); Study Completion 2023-02-03 (Estimated)

PRIMARY OUTCOMES:
Difference in percent of time spent with blood glucose level below 70 mg/dL | 3 months
  Baseline-treatment difference in % of time spent with blood glucose level below 70 mg/dL over the 3 months follow-up

SECONDARY OUTCOMES:
Percent of time within target range 70-180 mg/dL | 3 months
Percent of time spent with blood glucose level above 180 mg/dL | 3 months
Mean blood glucose level | 3 months
Percent of time spent with blood glucose level below 54 mg/dL | 3 months
Percent of time spent with blood glucose in range 70-140 mg/dL | 3 months
Glucose variability measured with the coefficient of variation (CV) | 3 months
Glucose variability measured with the standard deviation (SD) | 3 months
Percent of time spent with blood glucose level below 60 mg/dL | 3 months
Low blood glucose index (LBGI) | 3 months
  <2.5 low risk , [2.5-5] medium risk, >5 high risk
Hypoglycemia events (defined as at least 15 consecutive minutes <70 mg/dL) | 3 months
Percent of time spent with blood glucose level above 250 mg/dL | 3 months
Percent of time spent with blood glucose level above 300 mg/dL | 3 months
High blood glucose index (HBGI) | 3 months
  <2.5 low risk , [2.5-5] medium risk, >5 high risk
HbA1c at 3 months | at 3 months
HbA1c change from baseline to 3 months | 3 months
Fear of Hypoglycemia Survey | 3 months
  Total score from 0 (no fear) to 132 (important fear)
Hyperglycemia Avoidance Scale | 3 months
  Total score from 0 (do not avoid) to 40 (always avoid)
Diabetes Distress Scale | 3 months
  Total score range from 28 (low stress) to 168 (high stress)
Hypoglycemia Confidence Scale | 3 months
  Total score from 0 (no confidence) to 36 (very confident)
Clarke Hypoglycemia Awareness | 3 months
  Score range from 0 to 7. If more than 4 : reduced perception, if less : normal perception.
INSPIRE survey | 3 months
  Total score from 0 (high acceptance) to 110 (low acceptance)
System Usability Scale (SUS) | 3 months
  Total score from 0 (low acceptance) to 100 (high acceptance)
Insulin | 3 months
  Total daily insulin (units/kg), Basal: bolus insulin ratio
Weight and Body Mass Index (BMI) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric M RENARD, MD, PhD, Principal Investigator — Montpellier University Hospital
Locations (2):
- France (2):
  - University Hospital of Caen, Caen
  - UH Montpellier, Montpellier

IPD SHARING:
Plan to Share IPD: Yes
Sharing with NIDDK
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Renard E, Joubert M, Villard O, Dreves B, Reznik Y, Farret A, Place J, Breton MD, Kovatchev BP; iDCL Trial Research Group. Safety and Efficacy of Sustained Automated Insulin Delivery Compared With Sensor and Pump Therapy in Adults With Type 1 Diabetes at High Risk for Hypoglycemia: A Randomized Controlled Trial. Diabetes Care. 2023 Dec 1;46(12):2180-2187. doi: 10.2337/dc23-0685. PMID 37729080